CLINICAL TRIAL: NCT03131258
Title: The Effects of Pre-operative Anxiety on Anesthetic Recovery and Post-operative Pain in Donor Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, ERBIL TURKSAL, MD, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-5.1/5
Record Dates: First submitted 2017-02-10; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Kidney Transplantation; Anxiety; Pain, Acute; Anesthesia Recovery Period
MeSH Terms: conditions — Anxiety Disorders; Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Donor Nephrectomy (Other): Donor Nephrectomy
  Interventions: Procedure: Donor Nephrectomy

INTERVENTIONS:
Procedure: Donor Nephrectomy — 48 Donor Nephrectomy Patients

SUMMARY:
Kidney transplant is the most effective choice of treatment for patients with end-stage kidney failure in terms of quality of life and longevity. Today, 20-25% of kidney transplantations are implemented with living donors.

Donor nephrectomy is an operations which has the end goal of a living donor donating one of his kidneys to a patient with end-stage kidney failure (1).

Pre-operative anxiety is a condition which is characterized by a random illness, being hospitalised, anesthesia, surgery, or uneasiness or anxiety stemming from not knowing what is to be experienced. Educating and informing in the pre-operative period is the first step in mentally preparing the patient for the operation. In some studies, it has been pointed out that patients who were thoroughly informed in the pre-operative period have lower anxiety levels both in the pre-operative and post-operative periods with also less levels of pain and increased recovery rates in the latter (2).

Anesthetic recovery starts at the end of the surgical process and ends with the anesthetized patient completely regaining a wide-awake, responsive state, defensive reflex, and muscle strength.

Post-operative pain is acute pain which starts with surgical trauma and ends with tissue healing (3). Providing optimal post-operative analgesia plays an important role in the prevention of post-operative complications (1,4,5).

There are studies which examine the link between pre-operative anxiety and post-operative pain (59,74,74,77,78). Patients who will undergo a donor nephrectomy constitute a specific group of patients both because they are not operated due to a health problem that they have and because the operation results with them losing an organ. There are no prospective studies about the effects of pre-operative anxiety on anesthetic recovery and post-operative pain in individuals who have undergone donor nephrectomy in literature. Because of this, we have aimed to research prospectively the effects of pre-operative anxiety on anesthetic recovery and post-operative pain in patients that were to undergo donor nephrectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II between 18-60 years
* Donor Nephrectomy patients

Exclusion Criteria:

* psychiatric disturbance
* medicinal allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | 48 hours
  Patient's pain intensity as measured by visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Erbil Türksal, MD, Principal Investigator — Ege University

IPD SHARING:
Plan to Share IPD: Yes